# Age-related Macular Degeneration (AMD) in the Vitamin D and Omega-3 Trial (VITAL)

NCT01782352

(3/29/2012)

# Protocol: AMD in the VITamin D and OmegA-3 TriaL (VITAL)

(Version 1: 3/29/2012)

### I. BACKGROUND AND SIGNIFICANCE

Age-related macular degeneration (AMD) is the leading cause of blindness in the US. An estimated 1.75 million US men and women suffer from the advanced forms of geographic atrophy or neovascular AMD, and another 7 million are at substantial risk of this outcome. 1 Despite advances in photodynamic 2 and antivascular endothelial growth factor therapy<sup>3, 4</sup> for patients with neovascular AMD, and the demonstration of benefit from a supplement of antioxidants plus zinc for people with intermediate to advanced AMD,<sup>5</sup> vision loss from AMD remains commonplace. **VITAL-AMD** will use the resources of the **VIT**amin D and Omeg**A**-3 Tria**L** (**VITAL**) (U01 CA138962; JoAnn Manson, PI) to test the efficacy of two promising preventive agents in delaying the incidence and progression of AMD among 20.000 older men and women. Vitamin D3 and omega-3 fatty acids share anti-inflammatory, antioxidant, antiproliferative, and antiangiogenic properties, and evidence supports potential benefits of both agents as strong candidates for prevention of AMD. VITAL-**AMD** will have strong statistical power to address the primary (incidence) and secondary (progression to advanced stages) prevention of AMD. Findings from this study will clarify whether these agents reduce incidence and progression of AMD, and will provide important data for both public health and clinical guidelines for the primary and secondary prevention of AMD.

Role of DHA+EPA in AMD - Docosahexaenoic acid (DHA) and eicosapentaenoic acid (EPA) are marine omega-3 polyunsaturated fatty acids that can be synthesized from alpha-linolenic acid, though the major source is through diet. DHA and EPA are important in the developing eye and visual processing. DHA is found in neural and vascular cell membranes and is a major structural component of photoreceptor outer segments.<sup>6</sup> DHA is required for normal photoreceptor function,<sup>7</sup> and it accounts for the permeability and fluidity of outer segment membranes.<sup>8, 9</sup> DHA protects the vascular and neural retina from a range of stressors including reactive oxygen, ischemia, and inflammation, and helps promote survival of photoreceptor and RPE cells during phagocytosis.<sup>10</sup> The distal tips of photoreceptor outer segments are intermittently shed and renewed, necessitating a constant supply of DHA and EPA. DHA insufficiency is associated with a delay in photoreceptor response and alterations in retinal structure and function that could influence the onset and progression of AMD.<sup>11</sup> Supplementation with DHA and EPA appears to reverse these deficits<sup>12</sup> and could have a similar beneficial effect on AMD.

EPA is concentrated in the retinal vascular endothelium and in blood components<sup>13</sup> and has potent anti-inflammatory properties. EPA regulates lipoprotein metabolism and inhibits expression of several inflammatory mediators (e.g. intercellular adhesion molecule (ICAM)-1, monocyte chemotactic protein (MCP)-1, vascular endothelial growth factor (VEGF) and interleukin (IL)-6).<sup>14, 15</sup> EPA also inhibits nuclear factor κB (NF-κB) activation, and thus expression of a number of inflammatory compounds that can damage the Bruch membrane and lead to AMD.<sup>16</sup> NF-κB is a central regulator of IL-6, a critical regulator of CNV.<sup>15</sup> EPA is the precursor to a group of

eicosanoids (e.g. series-3 prostaglandins and series-5 leukotrienes) that counteract series-2 prostaglandins derived from arachidonic acid that promote inflammation, cell proliferation, and angiogenesis and interfere with immune cell function. <sup>13</sup> EPA and DHA also produce resolvins, which stop infiltration and transmigration of polymorphonuclear leukocytes, block the production of pro-inflammatory mediators and regulate the trafficking of leukocytes, cells and mediators to sites of inflammation. <sup>17</sup> Further, EPA depresses VEGF-specific tyrosine kinase receptor activation and expression, <sup>18</sup> and with DHA may reduce neovascularization independent of VEGF. <sup>19</sup> Recent work has shown that omega-3 fatty acids attenuate choroidal neovascularization in mice, <sup>15</sup> and reduce or reverse retinal lesions in the Ccl2-/-/Cx3cr1-/- mouse model of AMD. <sup>20</sup> Such findings are in line with epidemiological evidence in humans.

Some cross-sectional studies have reported significant inverse associations between higher fish intake and risk of early<sup>21</sup> or late AMD,<sup>22-26</sup> while others found no association.<sup>27-29</sup> Among studies examining omega-3 fatty acids, 2 studies found no significant relationships, 21, 30 whereas 4 studies showed reduced risks of neovascular AMD<sup>22-24</sup> or central geographic atrophy, <sup>25</sup> although in 2 studies the benefit was restricted to those with low dietary intake of linoleic acid. 22, 23 Prospective studies include a report on 567 incident cases of AMD from the Nurses' Health Study (NHS) and Health Professionals Follow-up Study (HPFS) that showed a significant 30% reduction in AMD incidence with high DHA intake (RR not significant after adjustment for other fats).31 High intake of EPA was associated with a non-significant 23% lower risk of AMD. In the Blue Mountains Eye Study, higher intake of omega-3 fatty acids lowered risk of early AMD by 60% after 5 y.32 At 10 y, the reduction was attenuated and not significant.<sup>33</sup> In the Melbourne Collaborative Cohort Study, higher omega-3 fatty acid intake reduced early AMD risk by 15%.34 In the Age-related Eye Disease Study (AREDS), after 6.3 y of follow-up, risks for central geographic atrophy were 45% & 56% lower in those with high intake of DHA & EPA, respectively.35 Higher intakes of DHA & EPA were also associated with ~25% lower risks for progression to advanced AMD after 8 y follow-up in AREDS.36 At 12 y, there continued to be a significant ~30% reduction in risk of advanced AMD for EPA & DHA,<sup>37</sup> as well as total intake of omega-3 fatty acids.<sup>38</sup> A meta-analysis showed that a high intake of omega-3 fatty acids conferred a 38% risk reduction for advanced AMD, and fish intake ≥2x/wk was associated with 25% and 33% lower risks of early and advanced AMD, respectively.<sup>39</sup>

We recently examined dietary intake of omega-3 fatty acids and AMD among 38,022 women in the Women's Health Study (WHS) who completed a dietary questionnaire at baseline and were free of a diagnosis of AMD. A total of 235 cases of visually significant AMD were confirmed during 10 y of follow-up. Women in the highest third of DHA intake had a 38% lower risk of AMD (RR, 0.62; 95% CI, 0.44-0.87) compared to those in the lowest third of intake. High intake of EPA was also associated with a reduced risk of AMD (RR, 0.66; 95% CI, 0.48-0.92). These prospective data from a large population of women appear to be the strongest evidence to date to support a role for DHA and EPA in the primary prevention of AMD.

Possible Mechanisms for Vitamin D in AMD - A plausible role for vitamin D3 in AMD prevention can be postulated due to its immunomodulatory, anti-inflammatory, and antiangiogenic properties. 1,25(OH)2D interferes with the activation and signaling of NF-κB.<sup>40, 41</sup> 1,25(OH)2D decreases production of proinflammatory cytokines IL-2,42 IL-6,43 IL-8,44 and IL-12,45 increases production of the antiinflammatory cytokine IL-10,46 and regulates expression of matrix metalloproteinase-9.47 Vitamin D also lowers blood levels of C-reactive protein, a marker of systemic inflammation that we have prospectively linked to elevated risks of AMD in the WHS<sup>48</sup> and others have shown to be associated with AMD.<sup>49-52</sup> Vitamin D is a potent stimulator of mechanisms for pathogen elimination, which could be relevant given the possible involvement of chronic infection in AMD.53 In addition, vitamin D regulates the renin-angiotensin-aldosterone system (RAAS) via suppression of renin gene expression and biosynthesis,54 and could exert an indirect beneficial effect on AMD through improved blood pressure control. 55 Favorable effects of vitamin D on glucose tolerance and insulin sensitivity<sup>56, 57</sup> could also mediate a beneficial effect in AMD as suggested by the association between dietary glycemic index and AMD. 58-62

In vitro and in vivo studies have demonstrated that 1,25(OH)2D profoundly inhibits growth of a variety of tumors by directly impacting the proliferation and activity of endothelial cells (ECs) and inhibiting angiogenesis, actions mediated by VDR.<sup>63-65</sup> In the mouse oxygen-induced ischemic retinopathy (OIR) model, 1,25(OH)2D-treated animals demonstrated a dose-dependent reduction in retinal neovascularization, and inhibition of retinal EC capillary morphogenesis without a significant inhibitory effect on EC proliferation and migration.<sup>66</sup>

To date, there are 3 studies of vitamin D and AMD, all supportive. Circulating 25(OH)D reflects all sources of vitamin D exposure, has a half-life of 2-3 weeks, and is the most comprehensive and stable indicator of vitamin D status.<sup>67</sup> Data from the 3rd NHANES indicated that serum levels of 25(OH) D were inversely associated with the prevalence of early AMD (OR for extreme quintiles, 0.64, 95%CI, 0.5-0.8), but not advanced AMD (OR, 1.16, 95%CI, 0.5-3.1).<sup>68</sup> Data from the Carotenoids and Age-Related Eye Disease Study indicated that high serum 25(OH)D status may be protective against intermediate AMD in women <75 y (OR for extreme quintiles, 0.57; 95% CI, 0.33-0.99; p=0.02).<sup>69</sup> Recent data from a monozygotic twin study with discordant AMD phenotypes found higher dietary intake of vitamin D in the twin with less severe AMD.<sup>70</sup>

#### II. SPECIFIC AIMS

The primary aims of this proposal are:

- 1. Does fish oil supplementation (EPA+DHA, 1g/d), compared to placebo, reduce the incidence and/or progression of AMD?
- 2. Does vitamin D3 supplementation (2000 IU/d), compared to placebo, reduce the incidence and/or progression of AMD?

The primary aims will be addressed in analyses involving the entire **VITAL** cohort of n=20,000 older men and women.

The secondary aims of this proposal are:

3. Are there synergistic or antagonistic effects of fish oil and vitamin D3 supplementation on the primary and secondary AMD endpoints?

This secondary aim will be addressed in analyses involving the entire *VITAL* cohort of n=20,000 older men and women.

- 4. Does baseline circulating vitamin D status modify the effect of vitamin D3 supplementation on AMD?
- 5. Does baseline circulating omega-3 fatty acid status modify the effect of EPA+DHA supplementation on AMD?

Secondary aims 4 and 5 will be addressed in the subgroup which provides a baseline blood specimen (N~16000).

- 6. Are there associations of polymorphisms in CYP24A1, vitamin D receptor, desaturase genes, or other genes with functional relevance to vitamin D and omega-3 fatty acid pathways with incidence of AMD?
- 7. Do polymorphisms in CYP24A1, the vitamin D receptor, complement factor H, ARMS2, C3, C2/BF, RORA, or other functionally relevant genes modify the effects of vitamin D3 on the AMD endpoints?
- 8. Do polymorphisms in desaturase genes (FADS1, FADS2, FADS3), elongase of very long fatty acids 2 (ELOVL2), complement factor H, ARMS2, C3, C2/BF, RORA, or other functionally relevant genes modify the effects of EPA+DHA on the AMD endpoints?

Secondary aims 6, 7, and 8 will be addressed in the subgroup which provides a baseline blood specimen using a nested case-control sample of all AMD cases (incident AMD cases and progression to advanced AMD) and a set of age- and sexmatched controls remaining free of AMD.

#### III. SUBJECT SELECTION/ENROLLMENT

**VITAL-AMD** is an ancillary study of the NIH-funded **VITAL** trial. All persons randomized in **VITAL** are included in this ancillary study.

Individuals are eligible for *VITAL* trial participation if they meet the following criteria: (1) are age ≥60 (men) or ≥65 (women); (2) have at least a high school education (to complete mail-based questionnaires); (3) have no history of cancer (except non-melanoma skin cancer), MI, stroke, TIA, angina pectoris, CABG, or PCI; (4) have none of the following safety exclusions: history of kidney stones, renal failure or dialysis, hypercalcemia, hypo-or hyperparathyroidism, severe liver disease (cirrhosis), or sarcoidosis or other granulomatous diseases such as active chronic tuberculosis or Wegener's granulomatosis; (5) have no allergy to fish (for EPA+DHA); (6) have no other serious illness that would preclude participation; (7)

are consuming no more than 800 IU of vitamin D from all supplemental sources combined (individual vitamin D supplements, calcium+vitamin D supplements, medications with vitamin D [e.g., Fosamax Plus D], and multivitamins), or, if taking, willing to decrease or forego such use during the trial (to ensure the overall dose is well below the no-observed-adverse effect level (NOAEL) of 4000 IU specified by the European Commission Scientific Committee on Food (ECSCF); (8) are consuming no more than 1200 mg/d of calcium (the RDA) from all supplemental sources combined, or, if taking, willing to decrease or forego such use during the trial; (9) are not taking fish oil supplements, or, if taking, willing to forego their use during the trial; and (10) are willing to participate, as evidenced by signing the informed consent form.

# IV. STUDY PROCEDURES

The procedures used to ascertain and document self-reports of AMD in *VITAL-AMD* are modeled on those used for more than two decades by the PIs in Physicians' Health Study I and II, Women's Health Study, and Women's Antioxidant Folic Acid Cardiovascular Study. All information is obtained masked to randomization status. Baseline and follow-up questionnaires are sent to study participants annually to obtain reports of diagnoses of AMD. Non-respondents are sent additional requests and are finally called to ensure complete follow-up. Reports of AMD may also be received through letters or telephone calls. Following the report of AMD, we obtain written consent to identify the diagnosing eye doctor(s) and obtain medical record information. We will contact the eye doctor(s) by mail and request they complete an AMD questionnaire or forward a complete copy of the patient's medical records pertaining to the diagnosis of AMD.

AMD questionnaire - The AMD questionnaire asks about the date of initial diagnosis of AMD, the best-corrected visual acuity (VA) at the time of diagnosis, the date when VA reached 20/30 or worse, the most recent VA, and information about the pathological findings observed on exam (drusen, RPE hypo- &/or hyperpigmentation, geographic atrophy, RPE detachment, subretinal neovascular membrane, or disciform scar). The questionnaire will inquire about drusen size (small, intermediate, large) as well as information on the location of geographic atrophy (central versus noncentral). We will obtain information on treatments for AMD (laser, photodynamic, or anti-VEGF therapy). We will also obtain information about whether there are other ocular abnormalities that could explain or contribute to visual loss. If so, the eye doctor is asked to provide his/her judgment as to whether AMD, by itself, is significant enough to cause VA of 20/30 or worse. Once obtained, the medical record information will be evaluated by a single reviewer (Dr. Christen), masked to the treatment assignments, to determine conformity with uniform diagnostic criteria. In cases of uncertainty, Dr. Schaumberg will also review the records. Reports for which doctors indicate diagnostic uncertainty will not be included as cases. When other ocular pathology is present, we will not include the case in our visually-significant AMD case group unless the examining eye doctor indicates their judgment that the AMD by itself would be sufficient to result in VA of 20/30 or worse. We define neovascular AMD by presence of RPE detachment, subretinal neovascular membrane, or disciform scar, either from clinical exam,

photos, or OCT if available, and will document the date of diagnosis of neovascular AMD.

Fundus Photographs - In order to obtain the highest quality endpoints possible in **VITAL-AMD**, we will obtain standard fundus photographs (e.g. 30° color photographs centered on the macula) of each eye from all participants for whom we confirm a diagnosis of AMD by review of medical records. In our recent experience, nearly all cases of neovascular AMD have photographs, angiograms, or OCTs available as part of routine care, however, dry AMD cases may not have photos. We will take the following steps to obtain photos for each prevalent case at baseline and for all incident cases: 1) When we obtain the medical record information, we will request copies of fundus photos centered on the macula for both eyes if available, or if not available we will ask whether the doctor would be willing and able to obtain a new set of photos for VITAL-AMD. 2) Study participants who do not already have photos in their medical records will be asked whether they would be willing to have photos taken (we have received funds to reimburse clinics for taking and sending photographs for VITAL participants with AMD), 3) If the participant's own doctor is not willing or able to take a set of photographs (e.g. s/he doesn't have the equipment), we will assist participants to obtain photographs from a doctor near their home. We will use databases (e.g. the Academy of Ophthalmology maintains a list by subspecialty) to search for retina specialists or other eye doctors with offices near the study participant and ascertain their willingness to take a set of photos for VITAL-AMD. 4) At the end of the trial, we will obtain a 2nd set of photos from all cases who remain alive and for whom we have not already documented progression to advanced AMD. 5) We will use the simplified AREDS scale to evaluate the photographs (grading will be done masked to randomization status).

Assessment of AMD progression. - We will send an annual follow-up questionnaire to all participants with medical-record confirmed AMD to ascertain progression to advanced AMD. The questionnaire will ask about changes in the participant's vision, and any updates on their diagnosis of AMD (e.g. the development of the "wet" form, any treatments received [e.g. anti-VEGF therapy], etc.). We will obtain follow-up medical records from all cases in which we suspect progression may have occurred. We will also routinely obtain follow-up records every two years from all participants with confirmed AMD that has not yet progressed to advanced AMD to help ensure no cases of progression are missed. Finally, we will also obtain a second set of retinal photographs at the end of the trial and grade these using the simplified AREDS scale. Progression along the simplified AREDS scale will be ascertained during analysis by comparison of the final grade with the baseline grade.

Validity of medical record-confirmed incident AMD - At initiation of VITAL-AMD we will conduct a pilot study to further validate our methodology for collection of photographs and to estimate sensitivity of case detection in the VITAL population. We will immediately seek to obtain informed consent for review of eye exam records and retinal photographs from a sample of 500 randomly selected VITAL participants at baseline. We will review medical records and photos masked to both randomized treatment assignments as well as the participants' response to the question about a prior diagnosis of AMD. We will estimate sensitivity based on the proportion of true

positives, that is the proportion of true AMD cases (identified by reviewing medical records and photos) that we identified using our methodology for AMD case identification (i.e. those that reported AMD on the baseline questionnaire that were confirmed by review of medical records). With estimated baseline prevalence of AMD=0.07 we will be able to estimate sensitivity with a 95% CI of ±15%. If sensitivity is found to be too low (e.g. <65%), we will consider strategies for increasing case detection in *VITAL-AMD*, for example by increasing participant awareness of AMD and the importance of eye exams for its detection, e.g. through participant newsletters.

#### V. BIOSTATISTICAL ANALYSIS

Assuming annual event rates for AMD observed in our previous trials of men and women, and an average follow-up of 6 years (expected for *VITAL*), *VITAL-AMD* will have good (≥80%) to excellent (≥95%) power to detect reductions of ≥20% in the primary AMD endpoint.

The study design is a 2x2 factorial randomized trial. With the large sample size, randomization should assure an equal distribution of known and unknown confounders between treatment groups, but we will control in analysis for any chance imbalances that may occur for AMD risk factors or conditions requiring more frequent medical attention that could increase the likelihood of AMD diagnosis. We will estimate the main treatment effects using the intention-to-treat principle based on randomized treatment assignment. Initial analyses of primary and secondary AMD endpoints will include contingency tables in which the rate of each endpoint (number of events per person-year of observation) among participants allocated to active treatment will be compared with the rate among those allocated to its placebo; controlling by stratification for the other treatment assignment. In addition, Kaplan-Meier survival estimates, the logrank test, and proportional hazards regression models201 will be used to determine whether there is a difference in time to an AMD event. Because an extended exposure to the study agents may be required to observe an effect, we will also conduct analyses which exclude AMD events that occur during the early years after randomization. To address the issue of AMD ascertainment, we will also test associations in models where the at-risk population during each 1 y follow-up period is restricted to those who report having had an eye exam during that year.

We will examine effect modification by the other randomized intervention, by race/skin pigmentation (for vitamin D), and by other risk factors by including an interaction term in proportional hazards models, as well as using methods for testing additive interactions. Stored blood samples will be used to measure genetic polymorphisms and analyses will examine the effect of these polymorphisms on the AMD endpoints, as well as modification of the treatment effects. These analyses will be analyzed as a nested case-control study using multivariable conditional logistic regression analyses and will also include testing of interactions on the additive scale.

#### VI. RISKS AND DISCOMFORTS

The only possible risk in this study involves the social/psychological risk that could result from inadvertent disclosure of confidential information from the questionnaires or blood tests. However, we have many safeguards in place to avoid this possibility, and we have never had an inadvertent breach of confidentiality in any of our trials. Confidentiality of participants is secured via locked file cabinets, use of participant ID numbers, and restrictions on access to computerized records and use or release of both individual and aggregate *VITAL* participant data, including randomized treatment assignments, in publications and presentations. Access to the *VITAL* databases and certain network files is restricted to essential staff only, and is protected by passwords and restricted access accounts. All blood specimens sent to the laboratories for analysis will be labeled with an ID number only, so that no individual identifying information will be made available in any form to these sites. In addition, employees involved with the proposed study will be asked to sign a form agreeing not to disclose any information to which they might have access, regardless of their personal perception about its confidentiality.

There is no additional risk to participation in **VITAL-AMD** beyond that incurred by participants as part of their regular activities in **VITAL**. All participants will have agreed by signing their **VITAL** consent form that their blood and other relevant data will be stored for future analyses and that they would not learn of the results of those analyses.

#### VII. POTENTIAL BENEFITS

For the majority of participants, there will be few direct benefits from participating in this primary prevention study other than the awareness of being involved in a large endeavor to answer relevant and timely questions regarding the possible benefits of vitamin D and marine omega-3 fatty acids. The potential benefits to society relate to the increasing use of both vitamin D and fish oil for many health purposes, with data not yet clearly indicating either clear benefit or harm. This study will provide a wealth of data on the effects of these supplements on risk of AMD, the leading cause of blindness in the United States, and will help guide individual decisions, clinical recommendations, and public health guidelines.

# VIII. MONITORING AND QUALITY ASSURANCE

As Co-Pls, Dr. William Christen and Dr. Debra Schaumberg will be responsible for monitoring data collection and assuring the validity and integrity of the data and adherence to the IRB-approved protocol.

A *VITAL* Data and Safety Monitoring Board (DSMB) has been created as an independent body charged with ensuring that the safety of participants is protected and that the scientific goals of the study are being met. The *VITAL* DSMB is charged with monitoring differences by treatment agent of ancillary study outcomes, including AMD, and will be empowered to terminate the trial based on evidence of substantial harm or benefit. To support those purposes, the DSMB will review any proposed amendments to the study protocol, examine the progress of the trial and the unblinded data on study endpoints, perform expedited review of all serious adverse

events (i.e., events meeting the FDA definition of Serious Adverse Events, such as any fatal event including suicide, immediately life-threatening event, or permanently or substantially disabling event), perform ongoing monitoring of drop-outs and nonserious adverse events, determine whether study procedures should be changed or the study should be halted for reasons related to the safety of participants, and perform periodic review of the completeness and validity of data to be used for analysis of safety and efficacy. The DSMB will also ensure participant privacy and research data confidentiality. The DSMB will employ monitoring rules<sup>71,72</sup> that will serve solely as guidelines in decisions regarding continuation or stopping of treatment arms. While these rules are intended for the primary endpoints of VITAL (primary prevention of cancer and CVD), the DSMB will also consider secondary and ancillary VITAL endpoints (including AMD) in assessing the overall balance of benefits and risks of the two agents. All decisions must be made after examining the totality of evidence, including other trial data, on these agents. All decisions will be made after examining the totality of evidence, including other trial data, on these agents.

### IX. REFERENCES

- 1. Friedman DS, O'Colmain BJ, Munoz B, et al. Prevalence of age-related macular degeneration in the United States. Arch Ophthalmol 2004;122(4):564-72.
- 2. Miller JW, Schmidt-Erfurth U, Sickenberg M, et al. Photodynamic therapy with verteporfin for choroidal neovascularization caused by age-related macular degeneration: results of a single treatment in a phase 1 and 2 study. Arch Ophthalmol 1999:117(9):1161-73.
- 3. Brown DM, Kaiser PK, Michels M, et al. Ranibizumab versus verteporfin for neovascular age-related macular degeneration. N Engl J Med 2006;355(14):1432-44.
- 4. Rosenfeld PJ, Brown DM, Heier JS, et al. Ranibizumab for neovascular agerelated macular degeneration. N Engl J Med 2006;355(14):1419-31.
- 5. A randomized, placebo-controlled, clinical trial of high-dose supplementation with vitamins C and E, beta carotene, and zinc for age-related macular degeneration and vision loss: AREDS report no. 8. Arch Ophthalmol 2001;119(10):1417-36.
- 6. Fliesler SJ, Anderson RE. Chemistry and metabolism of lipids in the vertebrate retina. Prog Lipid Res 1983;22(2):79-131.
- 7. Neuringer M, Anderson GJ, Connor WE. The essentiality of n-3 fatty acids for the development and function of the retina and brain. Annu Rev Nutr 1988;8:517-41.
- 8. Treen M, Uauy RD, Jameson DM, et al. Effect of docosahexaenoic acid on membrane fluidity and function in intact cultured Y-79 retinoblastoma cells. Arch Biochem Biophys 1992;294(2):564-70.
- 9. Niu SL, Mitchell DC, Litman BJ. Manipulation of cholesterol levels in rod disk membranes by methyl-beta-cyclodextrin: effects on receptor activation. J Biol Chem 2002;277(23):20139-45.
- 10. Mukherjee PK, Marcheselli VL, Serhan CN, Bazan NG. Neuroprotectin D1: a docosahexaenoic acid-derived docosatriene protects human retinal pigment epithelial cells from oxidative stress. Proc Natl Acad Sci U S A 2004;101(22):8491-6.
- 11. Hoffman DR, Birch DG. Docosahexaenoic acid in red blood cells of patients with X-linked retinitis pigmentosa. Invest Ophthalmol Vis Sci 1995;36(6):1009-18.
- 12. Anderson GJ, Neuringer M, Lin DS, Connor WE. Can prenatal N-3 fatty acid deficiency be completely reversed after birth? Effects on retinal and brain biochemistry and visual function in rhesus monkeys. Pediatr Res 2005;58(5):865-72.

- 13. SanGiovanni JP, Chew EY. The role of omega-3 long-chain polyunsaturated fatty acids in health and disease of the retina. Prog Retin Eye Res 2005;24(1):87-138.
- 14. Miles EA, Wallace FA, Calder PC. Dietary fish oil reduces intercellular adhesion molecule 1 and scavenger receptor expression on murine macrophages. Atherosclerosis 2000;152(1):43-50.
- 15. Koto T, Nagai N, Mochimaru H, et al. Eicosapentaenoic acid is anti-inflammatory in preventing choroidal neovascularization in mice. Invest Ophthalmol Vis Sci 2007;48(9):4328-34.
- 16. Chung HY, Cesari M, Anton S, et al. Molecular inflammation: underpinnings of aging and age-related diseases. Ageing Res Rev 2009;8(1):18-30.
- 17. Serhan CN. Systems approach with inflammatory exudates uncovers novel antiinflammatory and pro-resolving mediators. Prostaglandins Leukot Essent Fatty Acids 2008;79(3-5):157-63.
- 18. Yang SP, Morita I, Murota SI. Eicosapentaenoic acid attenuates vascular endothelial growth factor-induced proliferation via inhibiting Flk-1 receptor expression in bovine carotid artery endothelial cells. J Cell Physiol 1998;176(2):342-9.
- 19. Connor KM, SanGiovanni JP, Lofqvist C, et al. Increased dietary intake of omega-3-polyunsaturated fatty acids reduces pathological retinal angiogenesis. Nat Med 2007;13(7):868-73.
- 20. Tuo J, Ross RJ, Herzlich AA, et al. A high omega-3 fatty acid diet reduces retinal lesions in a murine model of macular degeneration. Am J Pathol 2009;175(2):799-807.
- 21. Delcourt C, Carriere I, Cristol JP, et al. Dietary fat and the risk of age-related maculopathy: the POLANUT study. Eur J Clin Nutr 2007;61(11):1341-4.
- 22. Seddon JM, Rosner B, Sperduto RD, et al. Dietary fat and risk for advanced agerelated macular degeneration. Arch Ophthalmol 2001;119(8):1191-9.
- 23. Seddon JM, George S, Rosner B. Cigarette smoking, fish consumption, omega-3 fatty acid intake, and associations with age-related macular degeneration: the US Twin Study of Age-Related Macular Degeneration. Arch Ophthalmol 2006;124(7):995-1001.
- 24. Augood C, Chakravarthy U, Young I, et al. Oily fish consumption, dietary docosahexaenoic acid and eicosapentaenoic acid intakes, and associations with neovascular age-related macular degeneration. Am J Clin Nutr 2008;88(2):398-406.
- 25. SanGiovanni JP, Chew EY, Clemons TE, et al. The relationship of dietary lipid intake and age-related macular degeneration in a case-control study: AREDS Report No. 20. Arch Ophthalmol 2007;125(5):671-9.
- 26. Swenor BK, Bressler S, Caulfield L, West SK. The impact of fish and shellfish consumption on age-related macular degeneration. Ophthalmology;117(12):2395-401.
- 27. Mares-Perlman JA, Brady WE, Klein R, et al. Dietary fat and age-related maculopathy. Arch Ophthalmol 1995;113(6):743-8.
- 28. Smith W, Mitchell P, Leeder SR. Dietary fat and fish intake and age-related maculopathy. Arch Ophthalmol 2000;118(3):401-4.
- 29. Heuberger RA, Mares-Perlman JA, Klein R, et al. Relationship of dietary fat to age-related maculopathy in the Third National Health and Nutrition Examination Survey. Arch Ophthalmol 2001;119(12):1833-8.
- 30. Sanders TA, Haines AP, Wormald R, et al. Essential fatty acids, plasma cholesterol, and fat-soluble vitamins in subjects with age-related maculopathy and matched control subjects. Am J Clin Nutr 1993;57(3):428-33.
- 31. Cho E, Hung S, Willett WC, et al. Prospective study of dietary fat and the risk of age-related macular degeneration. Am J Clin Nutr 2001;73(2):209-18.
- 32. Chua B, Flood V, Rochtchina E, et al. Dietary fatty acids and the 5-year incidence of age-related maculopathy. Arch Ophthalmol 2006;124(7):981-6.

- 33. Tan JS, Wang JJ, Flood V, Mitchell P. Dietary fatty acids and the 10-year incidence of age-related macular degeneration: the Blue Mountains Eye Study. Arch Ophthalmol 2009;127(5):656-65.
- 34. Chong EW, Robman LD, Simpson JA, et al. Fat consumption and its association with age-related macular degeneration. Arch Ophthalmol 2009;127(5):674-80.
- 35. SanGiovanni JP, Chew EY, Agron E, et al. The relationship of dietary omega-3 long-chain polyunsaturated fatty acid intake with incident age-related macular degeneration: AREDS report no. 23. Arch Ophthalmol 2008;126(9):1274-9.
- 36. Chiu CJ, Klein R, Milton RC, et al. Does eating particular diets alter the risk of age-related macular degeneration in users of the Age-Related Eye Disease Study supplements? Br J Ophthalmol 2009;93(9):1241-6.
- 37. SanGiovanni JP, Agron E, Clemons TE, Chew EY. Omega-3 long-chain polyunsaturated fatty acid intake inversely associated with 12-year progression to advanced age-related macular degeneration. Arch Ophthalmol 2009;127(1):110-2.
- 38. Sangiovanni JP, Agron E, Meleth AD, et al. {omega}-3 Long-chain polyunsaturated fatty acid intake and 12-y incidence of neovascular age-related macular degeneration and central geographic atrophy: AREDS report 30, a prospective cohort study from the Age-Related Eye Disease Study. Am J Clin Nutr 2009;90(6):1601-7.
- 39. Chong EW, Kreis AJ, Wong TY, et al. Dietary omega-3 fatty acid and fish intake in the primary prevention of age-related macular degeneration: a systematic review and meta-analysis. Arch Ophthalmol 2008;126(6):826-33.
- 40. McCarty MF. Targeting multiple signaling pathways as a strategy for managing prostate cancer: multifocal signal modulation therapy. Integr Cancer Ther 2004;3(4):349-80.
- 41. Janjetovic Z, Zmijewski MA, Tuckey RC, et al. 20-Hydroxycholecalciferol, product of vitamin D3 hydroxylation by P450scc, decreases NF-kappaB activity by increasing lkappaB alpha levels in human keratinocytes. PLoS One 2009;4(6):e5988.
- 42. Bemiss CJ, Mahon BD, Henry A, et al. Interleukin-2 is one of the targets of 1,25-dihydroxyvitamin D3 in the immune system. Arch Biochem Biophys 2002;402(2):249-54.
- 43. Sun X, Zemel MB. Calcitriol and calcium regulate cytokine production and adipocyte-macrophage cross-talk. J Nutr Biochem 2008;19(6):392-9.
- 44. Takahashi K, Horiuchi H, Ohta T, et al. 1 alpha,25-dihydroxyvitamin D3 suppresses interleukin-1beta-induced interleukin-8 production in human whole blood: an involvement of erythrocytes in the inhibition. Immunopharmacol Immunotoxicol 2002;24(1):1-15.
- 45. D'Ambrosio D, Cippitelli M, Cocciolo MG, et al. Inhibition of IL-12 production by 1,25-dihydroxyvitamin D3. Involvement of NF-kappaB downregulation in transcriptional repression of the p40 gene. J Clin Invest 1998;101(1):252-62.
- 46. Canning MO, Grotenhuis K, de Wit H, et al. 1-alpha,25-Dihydroxyvitamin D3 (1,25(OH)(2)D(3)) hampers the maturation of fully active immature dendritic cells from monocytes. Eur J Endocrinol 2001;145(3):351-7.
- 47. Timms PM, Mannan N, Hitman GA, et al. Circulating MMP9, vitamin D and variation in the TIMP-1 response with VDR genotype: mechanisms for inflammatory damage in chronic disorders? Qjm 2002;95(12):787-96.
- 48. Schaumberg DA, Christen WG, Buring JE, et al. High-sensitivity C-reactive protein, other markers of inflammation, and the incidence of macular degeneration in women. Arch Ophthalmol 2007;125(3):300-5.
- 49. Seddon JM, Gensler G, Milton RC, et al. Association between C-reactive protein and age-related macular degeneration. Jama 2004;291(6):704-10.

- 50. Seddon JM, George S, Rosner B, Rifai N. Progression of age-related macular degeneration: prospective assessment of C-reactive protein, interleukin 6, and other cardiovascular biomarkers. Arch Ophthalmol 2005;123(6):774-82.
- 51. Boekhoorn SS, Vingerling JR, Witteman JC, et al. C-reactive protein level and risk of aging macula disorder: The Rotterdam Study. Arch Ophthalmol 2007;125(10):1396-401.
- 52. Kikuchi M, Nakamura M, Ishikawa K, et al. Elevated C-reactive protein levels in patients with polypoidal choroidal vasculopathy and patients with neovascular agerelated macular degeneration. Ophthalmology 2007;114(9):1722-7.
- 53. Baird PN, Robman LD, Richardson AJ, et al. Gene-environment interaction in progression of AMD: the CFH gene, smoking and exposure to chronic infection. Hum Mol Genet 2008;17(9):1299-305.
- 54. Li YC, Kong J, Wei M, et al. 1,25-Dihydroxyvitamin D(3) is a negative endocrine regulator of the renin-angiotensin system. J Clin Invest 2002;110(2):229-38.
- 55. Weber KT, Simpson RU, Carbone LD. Vitamin D and calcium dyshomoeostasis-associated heart failure. Heart 2008;94(5):540-1.
- 56. Pittas AG, Harris SS, Stark PC, Dawson-Hughes B. The effects of calcium and vitamin D supplementation on blood glucose and markers of inflammation in nondiabetic adults. Diabetes Care 2007;30(4):980-6.
- 57. Mattila C, Knekt P, Mannisto S, et al. Serum 25-hydroxyvitamin D concentration and subsequent risk of type 2 diabetes. Diabetes Care 2007;30(10):2569-70.
- 58. Chiu CJ, Hubbard LD, Armstrong J, et al. Dietary glycemic index and carbohydrate in relation to early age-related macular degeneration. Am J Clin Nutr 2006;83(4):880-6.
- 59. Chiu CJ, Milton RC, Gensler G, Taylor A. Association between dietary glycemic index and age-related macular degeneration in nondiabetic participants in the Age-Related Eye Disease Study. Am J Clin Nutr 2007;86(1):180-8.
- 60. Chiu CJ, Milton RC, Klein R, et al. Dietary carbohydrate and the progression of age-related macular degeneration: a prospective study from the Age-Related Eye Disease Study. Am J Clin Nutr 2007;86(4):1210-8.
- 61. Kaushik S, Wang JJ, Flood V, et al. Dietary glycemic index and the risk of agerelated macular degeneration. Am J Clin Nutr 2008;88(4):1104-10.
- 62. Chiu CJ, Milton RC, Klein R, et al. Dietary compound score and risk of agerelated macular degeneration in the age-related eye disease study. Ophthalmology 2009;116(5):939-46.
- 63. Mantell DJ, Owens PE, Bundred NJ, et al. 1 alpha,25-dihydroxyvitamin D(3) inhibits angiogenesis in vitro and in vivo. Circ Res 2000;87(3):214-20.
- 64. Shokravi MT, Marcus DM, Alroy J, et al. Vitamin D inhibits angiogenesis in transgenic murine retinoblastoma. Invest Ophthalmol Vis Sci 1995;36(1):83-7.
- 65. Chung I, Han G, Seshadri M, et al. Role of vitamin D receptor in the antiproliferative effects of calcitriol in tumor-derived endothelial cells and tumor angiogenesis in vivo. Cancer Res 2009;69(3):967-75.
- 66. Albert DM, Scheef EA, Wang S, et al. Calcitriol is a potent inhibitor of retinal neovascularization. Invest Ophthalmol Vis Sci 2007;48(5):2327-34.
- 67. Giovannucci E. The epidemiology of vitamin D and cancer incidence and mortality: a review (United States). Cancer Causes Control 2005;16(2):83-95.
- 68. Parekh N, Chappell RJ, Millen AE, et al. Association between vitamin D and agerelated macular degeneration in the Third National Health and Nutrition Examination Survey, 1988 through 1994. Arch Ophthalmol 2007;125(5):661-9.
- 69. Millen AE, Voland R, Sondel SA, et al. Vitamin D status and early age-related macular degeneration in postmenopausal women. Arch Ophthalmol;129(4):481-9.

- 70. Seddon JM, Reynolds R, Shah HR, Rosner B. Smoking, dietary betaine, methionine, and vitamin D in monozygotic twins with discordant macular degeneration: epigenetic implications. Ophthalmology;118(7):1386-94.
- 71. Haybittle JL. Repeated assessment of results in clinical trials of cancer treatment. Br J Radiol 1971;44(526):793-7.
- 72. Peto R, Pike MC, Armitage P, et al. Design and analysis of randomized clinical trials requiring prolonged observation of each patient. I. Introduction and design. Br J Cancer 1976;34(6):585-612.